CLINICAL TRIAL: NCT02432469
Title: Quality Measurement and Improvement Study of Surgical Coronary Revascularization: Medication Adherence
Acronym: MISSION-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOST-2013BAI09B01-3
Record Dates: First submitted 2015-04-25; First posted 2015-05-04 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Bypass Grafting; Medication Adherence; Mobile Applications
Keywords: coronary artery bypass; medication adherence; secondary prevention; mobile applications
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): APP specific for this study, with reminder, education materials and feedback mechanism for improving secondary medications
  Interventions: Behavioral: APP intervention
- Control group (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: APP intervention — The APP contains education materials about secondary intervention of coronary artery disease, patients can surf and read them very easily. The APP also collects information on medication prescription by doctors, reminds patients at every time of taking medications, and asks for feedback from patients at 8 pm every day. The APP also pushes a patient-specific questionnaire with 10-15 questions weekly, to collect information about patients' medication adherence and self-management on blood pressure, blood lipid, blood glucose, physical activity, diet and body weight. APP pushes series of recommendations right after patients' finishing the questionnaire to help them improve their secondary prevention.
  Arms: Intervention group

SUMMARY:
The study is a randomized controlled trial, having a plan to recruit 1000 patients underwent coronary artery bypass grafting in 1 of 5 participating sites in 2015, and randomized to either the intervention group or control group, to test the effectiveness of a smartphone based application (APP) focusing on improving patients medication adherence. Patients randomized to the intervention group install the APP in their smartphones with personnel information and physicians' medication descriptions. The APP reminds at the time of taking medications, educates them on secondary prevention for coronary artery disease, and collects their weekly situations by questionaires. Investigators will follow-up patients by face to face or telephone interview. The 6-month effects of the intervention are evaluated.

DETAILED DESCRIPTION:
The aim of this study is to test the effectiveness of a smartphone based application (APP) on improvement of patients' adherence to medications after coronary artery bypass grafting.

DESIGN AND PROCEDURES The study is a randomized controlled trial, having a plan to recruit 1000 patients underwent coronary artery bypass grafting in 2015, and randomized to either the intervention group or the control group, to test the effectiveness of a smartphone based APP focusing on improving patients medication adherence. Patients randomized to the intervention group install the APP and are intervened by it. The patients randomized to control group receive usual care. The investigators follow up patients in both groups by face to face or telephone interview at 3-month and 6-month after randomization. The 6-month effects of the intervention are evaluated.

The APP contains education materials about secondary prevention of coronary artery disease, patients can surf and read easily. The APP also collects information on medication prescription by doctors, reminds patients at every time of taking medications, and asks for feedback at 8 pm everyday. The APP also pushes one patient-specific questionnaire with 10-15 questions weekly, to collect information about patients' medication adherence and self-administration on blood pressure, blood lipid, glucose, physical activity, diet and body weight. APP will push series of recommendations right after patients' finishing the questionnaire to help them improve secondary prevention.

The coordinators from participating sites interview patients at the baseline, 3-month and 6-month after the randomization, for information of medication adherence, major events and outcomes after coronary artery bypass grafting and quality of life. The primary outcome measure is the Chinese version of the 8-item Morisky medication adherence scale which has already been validated in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Underwent coronary artery bypass grafting in 2015

Exclusion Criteria:

* Does not use a smartphone
* Can not install the study specific APP into his/her smartphone
* Does not use 3 or more applications installed in his/her smartphone
* Is incapable to understand texts in Chinese
* Can not type numbers in his/her smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Medication adherence measured by Chinese version of the 8-item Morisky medication adherence scale (C-MMAC-8) | 6 months
  patients' medication adherence measured by C-MMAC-8 at 6-month after randomization, the scale of more than 7 is defined as adherence to medications

SECONDARY OUTCOMES:
Medication adherence measured by C-MMAC-8 | 3 month
  patients' medication adherence measured by C-MMAC-8 at 3-month after randomization, the scale of more than 7 is defined as adherence to medications
mortality at 6-month | 6 months
mortality at 3-month | 3 months
rate of major adverse cardiovascular or cerebral events at 6-month | 6 months
  composite endpoint of all-cause death, myocardial infraction, stroke and repeat revascularization
rate of major adverse cardiovascular or cerebral events at 3-month | 3 months
  composite endpoint of all-cause death, myocardial infraction, stroke and repeat revascularization

OTHER OUTCOMES:
pill count | 6 months
  the number of tablets remaining divided by the number of tablets prescribed
pill count | 3 month
  the number of tablets remaining divided by the number of tablets prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, MD, PhD, Study Director — State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, People's Republic of China; Zhe Zheng, MD, PhD, Principal Investigator — State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, People's Republic of China
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Yan J, You LM, Yang Q, Liu B, Jin S, Zhou J, Lin C, Morisky DE. Translation and validation of a Chinese version of the 8-item Morisky medication adherence scale in myocardial infarction patients. J Eval Clin Pract. 2014 Aug;20(4):311-7. doi: 10.1111/jep.12125. Epub 2014 May 10. PMID 24813538
- [Derived] Yu C, Liu C, Du J, Liu H, Zhang H, Zhao Y, Yang L, Li X, Li J, Wang J, Wang H, Liu Z, Rao C, Zheng Z; MISSION-2 Collaborative Group. Smartphone-based application to improve medication adherence in patients after surgical coronary revascularization. Am Heart J. 2020 Oct;228:17-26. doi: 10.1016/j.ahj.2020.06.019. Epub 2020 Jul 4. PMID 32745732
- [Derived] Liu CY, Du JZ, Rao CF, Zhang H, Liu HN, Zhao Y, Yang LM, Li X, Li J, Wang J, Wang HS, Liu ZG, Cheng ZY, Zheng Z. Quality Measurement and Improvement Study of Surgical Coronary Revascularization: Medication Adherence (MISSION-2). Chin Med J (Engl). 2018 Jun 20;131(12):1480-1489. doi: 10.4103/0366-6999.233767. PMID 29873315